CLINICAL TRIAL: NCT06368895
Title: Efficacy and Safety of Fecal Microbiota Transplantation by Oral Capsules in Patients With Liver
Brief Title: Fecal Microbiota Transplantation by Oral Capsules for Hepatic Encephalopathy Treatment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2188
Record Dates: First submitted 2024-04-04; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Hepatic Encephalopathy; Dysbiosis
MeSH Terms: conditions — Hepatic Encephalopathy; Dysbiosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fecal microbiota transplantation through colonoscopy and oral capsules (Experimental): Patients with cirrhosis and hepatic encephalopathy refractory to conventional treatment will undergo a two-stage fecal microbiota transplantation: initial colonoscopic delivery followed by daily oral capsules administration one month later. Patients will continue also conventional therapy with rifaximin and lactulose
  Interventions: Procedure: Fecal microbiota transplantation delivery through colonoscopy; Drug: Fecal microbiota transplantation delivery through oral capsules
- Fecal microbiota transplantation through oral capsules (Experimental): Patients with cirrhosis and hepatic encephalopathy refractory to conventional treatment will undergo fecal microbiota transplantation through daily oral capsules administration. Patients will continue also conventional therapy with rifaximin and lactulose.
  Interventions: Drug: Fecal microbiota transplantation delivery through oral capsules
- Controls (No Intervention): Patients with cirrhosis and hepatic encephalopathy refractory to conventional treatment will continue only conventional therapy with rifaximin and lactulose

INTERVENTIONS:
Procedure: Fecal microbiota transplantation delivery through colonoscopy — Patients will receive 4 L of macrogol and salts solution the afternoon before FMT and remain fasting the night before the scheduled treatment. During colonoscopy, about 350 mL of donor fecal preparation will be infused in the cecum.
  Arms: Fecal microbiota transplantation through colonoscopy and oral capsules
Drug: Fecal microbiota transplantation delivery through oral capsules — Intestinal gastro-resistant capsules (capacity 0.91 mL, overall 10^8-9 bacteria per capsule) will be filled with the fecal slurry. From each donation weighing 100 g, it is expected to obtain 150 cps, which will be promptly frozen and stored at -80°C. At each monthly visit, the patient will receive 60 capsules, to be stored at -20°C at home. Capsules will be administered orally at the dose of 1 cps twice a day from month 1 post-colonoscopy to patients in the FMT group 1 (colonoscopy plus capsules), and from day 1 to patients in the FMT group 2 (capsules only).
  Arms: Fecal microbiota transplantation through colonoscopy and oral capsules; Fecal microbiota transplantation through oral capsules

SUMMARY:
This interventional study aims to evaluate the safety and efficacy of oral capsule fecal microbiota transplantation (FMT) for treating hepatic encephalopathy refractory to conventional rifaximin and lactulose therapy in patients with liver cirrhosis. Patients diagnosed with hepatic encephalopathy refractory to rifaximin and lactulose therapy will be randomized into three groups. While continuing conventional therapy, the first group receives FMT via colonoscopy and oral capsule administration, the second group receives only oral capsule administration, and the third group serves as a control, receiving only conventional therapy.

The aims of the study are:

To evaluate the efficacy and safety of FMT by oral capsules in cirrhotic patients with hepatic encephalopathy refractory to standard therapy.

To evaluate changes in the gut microbiota composition and in the intestinal and systemic inflammatory condition occurring after FMT and if they can be associated with clinical improvement.

To evaluate metabolic modifications occurring after FMT and if they can be associated with clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of liver cirrhosis
* Hepatic encephalopathy of grade >1 or higher according to West Haven classification, persistent or recurrent despite treatment with lactulose/lactitol and rifaximin at adequate doses started at least 30 days before the Hepatic encephalopathy episode

Exclusion Criteria:

* Na <130 meq /l
* Creatinine > 1.3 mg / dl
* Presence of grade 3 ascites
* Presence of esophagogastric varices at risk of haemorrhage in the absence of adequate prophylaxis
* Presence of other possible causes of encephalopathy (cerebral vascular disease, known neurodegenerative or cognitive disorders)
* Known psychiatric disorders or other causes of brain dysfunction (e.g. hypoglycemia, hyponatremia)
* Alcohol consumption
* Diagnosis of hepatocellular carcinoma
* Contraindication to fecal microbiota transplantation (e.g. pregnancy or breastfeeding)
* Presence of known intestinal diseases
* Any clinical condition that, in the opinion of the investigators, may contraindicate the enrollment in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety of fecal microbiota transplantation by oral capsules in the treatment of cirrhotic patients with hepatic encephalopathy refractory to conventional therapy | 12 months
  Number of patients with treatment associated adverse events as assessed by CTCAE v5.0
Evaluation of efficacy of fecal microbiota transplantation by oral capsules in the treatment of cirrhotic patients with hepatic encephalopathy refractory to conventional therapy | 12 months
  Number of patients with an improvement or no worsening of hepatic encephalopathy after treatment administration as clinically assessed by West-Haven classification and psychometric tests (portosystemic hepatic encephalopathy syndrome test and inhibitory control test) and through laboratory measurement of ammonia serum levels.

SECONDARY OUTCOMES:
Evaluation of changes in the gut microbiota composition following the fecal microbiota transplantation | 12 months
  DNA and RNA microbiota sequencing on fecal samples will be performed every three months after treatment initiation to define changes in the abundance of bacteria and alpha diversity (by the Simpson's Index of Diversity).
Evaluation of changes in the systemic inflammatory following the fecal microbiota transplantation | 12 months
  Changes in the systemic inflammatory condition will be assessed by the quantification of serum cytokines, chemokines, and bacterial fragments concentrations (units/ml): Interleukin1 beta, tumor necrosis factor alpha, Interleukin2, Interleukin6, Interleukin17, interferon gamma, Chemokine C-C motif ligand 2, Chemokine C-C motif ligand 3, Chemokine C-C motif ligand 4, Chemokine C-C motif ligand 5, Chemokine C-C motif ligand 10, Chemokine C-X-C motif ligand 10, lipopolysaccharides
Evaluation of changes in the intestinal inflammatory following the fecal microbiota transplantation | 12 months
  Changes in the intestinal inflammatory condition will be assessed by the quantification of fecal calprotectin concentration (mg/dl).
Comparison between protein metabolites concentration (ppm) in serum, urine and feces before and after microbiota transplantation | 12 months
  Quantification of amino acides will be performed before the microbiota transplantation and every three months after by the examination of serum, urine and fecal samples through liquid chromatography tandem mass spectrometry methods.
Comparison between lipid metabolites concentration (ppm) in serum, urine and feces before and after microbiota transplantation | 12 months
  Quantification of fatty acids, acyl carnitine, tryglicerides, dyacil glycerols and phospholipides will be performed before the microbiota transplantation and every three months after by the examination of serum, urine and fecal samples through liquid chromatography tandem mass spectrometry methods.
Comparison between carbohydrates metabolites concentration (ppm) in serum, urine and feces before and after microbiota transplantation | 12 months
  Quantification of tricarboxylic acid cycle compounds, sugars and sugar phosphates will be performed before the microbiota transplantation and every three months after by the examination of serum, urine and fecal samples through liquid chromatography tandem mass spectrometry methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grover VP, Tognarelli JM, Massie N, Crossey MM, Cook NA, Taylor-Robinson SD. The why and wherefore of hepatic encephalopathy. Int J Gen Med. 2015 Dec 16;8:381-90. doi: 10.2147/IJGM.S86854. eCollection 2015. PMID 26719720
- [Background] American Association for the Study of Liver Diseases; European Association for the Study of the Liver. Hepatic encephalopathy in chronic liver disease: 2014 practice guideline by the European Association for the Study of the Liver and the American Association for the Study of Liver Diseases. J Hepatol. 2014 Sep;61(3):642-59. doi: 10.1016/j.jhep.2014.05.042. Epub 2014 Jul 8. No abstract available. PMID 25015420
- [Background] Bajaj JS, Hafeezullah M, Hoffmann RG, Saeian K. Minimal hepatic encephalopathy: a vehicle for accidents and traffic violations. Am J Gastroenterol. 2007 Sep;102(9):1903-9. doi: 10.1111/j.1572-0241.2007.01424.x. Epub 2007 Jul 19. PMID 17640323
- [Background] Fujisaka S, Avila-Pacheco J, Soto M, Kostic A, Dreyfuss JM, Pan H, Ussar S, Altindis E, Li N, Bry L, Clish CB, Kahn CR. Diet, Genetics, and the Gut Microbiome Drive Dynamic Changes in Plasma Metabolites. Cell Rep. 2018 Mar 13;22(11):3072-3086. doi: 10.1016/j.celrep.2018.02.060. PMID 29539432
- [Background] Bajaj JS. The role of microbiota in hepatic encephalopathy. Gut Microbes. 2014 May-Jun;5(3):397-403. doi: 10.4161/gmic.28684. Epub 2014 Apr 1. PMID 24690956
- [Background] Claesson MJ, Clooney AG, O'Toole PW. A clinician's guide to microbiome analysis. Nat Rev Gastroenterol Hepatol. 2017 Oct;14(10):585-595. doi: 10.1038/nrgastro.2017.97. Epub 2017 Aug 9. PMID 28790452
- [Background] Kelly CR, Kahn S, Kashyap P, Laine L, Rubin D, Atreja A, Moore T, Wu G. Update on Fecal Microbiota Transplantation 2015: Indications, Methodologies, Mechanisms, and Outlook. Gastroenterology. 2015 Jul;149(1):223-37. doi: 10.1053/j.gastro.2015.05.008. Epub 2015 May 15. PMID 25982290